CLINICAL TRIAL: NCT01918787
Title: Examine the Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) Over the Symptoms of Autism Spectrum Disorder
Brief Title: rTMS for Adults With Autistic Spectrum Disorder
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100-2985C; NSC 100-2314-B-182A-075 (Other: National Science Council)
Record Dates: First submitted 2013-08-02; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2012-04

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- repetitive TMS (Experimental): repetitive TMS over dorsolateral prefrontal cortex, posterior superior temporal sulcus and inion as control
  Interventions: Device: repetitive TMS

INTERVENTIONS:
Device: repetitive TMS — rTMS (intermittent theta burst stimulation 1200)over posterior superior temporal sulcus,dorsolateral prefrontal cortex and inion as Sham control

SUMMARY:
rTMS over dorsolateral prefrontal cortex is effective in reducing repetitive behaviors in adults with autistic spectrum disorder rTMS over posterior superior temporal sulcus is effective in improving social ability in adults with autistic spectrum disorder

DETAILED DESCRIPTION:
First, we will apply one session intermittent theta burst stimulation over dorsolateral prefrontal cortex, posterior superior temporal sulcus and inion as control with one week interval in adults with autism spectrum disorder. Second, we will apply 5 sessions intermittent theta burst stimulation within one week over dorsolateral prefrontal cortex or posterior temporal sulcus depending on the results of our first phases.

ELIGIBILITY:
Inclusion Criteria:

* adults with autistic spectrum disorder

Exclusion Criteria:

* schizophrenia
* bipolar affective disorder
* major depressive disorder
* any systemic disease especially epilepsy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
continuous performance test | continuous performance test will be arranged before and after rTMS within one hour
  continuous performance test will be arranged before and after rTMS within one hour

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | Yale-Brown Obsessive Compulsive Scale will be evaluated before and after rTMS within one week
  Yale-Brown Obsessive Compulsive Scale will be evaluated before and after rTMS. The time point of evaluation is before rTMS, one hour after rTMS, 3 days after rTMS and one week after rTMS.

OTHER OUTCOMES:
Autism Spectrum Quotient | Autism Spectrum Quotient will be evaluated before and after rTMS within one week
  Autism Spectrum Quotient will be evaluated before and after rTMS. The time point of evaluation is before rTMS, one hour after rTMS, 3 days after rTMS and one week after rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Chang Ni, MD, Principal Investigator — Chang Gung Memorial Hospital at Linkou, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan